CLINICAL TRIAL: NCT02130544
Title: Acute Pain Management Following Video-assisted Thoracoscopic Surgery: Comparison of Lobectomy and Wedge Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201403039RIND
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Viedo-assisted thoracoscopic surgery(VATS) have became popular in recent years. There is no golden rule of postoperative analgesia for VATS. Compared with lobectomy, wedge resection preserves better pulmonary function and is suitable for elder patients and patients who could not afford to have lobectomy. In addition to surgery time、recovery time and hospital stay, wound incisions and organization damages are different,too. Will patients also have different response to pain control after these two surgery? The retrospective study is to compared the differences of postoperative pain management between VATS lobectomy and wedge resection.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 20
2. Using intravenous patient-controlled analgesia for postoperative analgesia
3. ASA physical status classification I-III

Exclusion Criteria:

1. Staying in intensive care unit after surgery
2. Emergency surgery
3. Pregnancy
4. Other surgery incisions which are not used for the video-assisted thoracoscopic surgery
5. Patients never use intravenous patient-controlled analgesia after surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Selected patients are from the hospital patients who are arranged to have video-assisted thoracoscopic surgery for lobectomy or wedge resection
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain scale | postoperative day 1 to day 3

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Jung Cheng, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan